CLINICAL TRIAL: NCT00743405
Title: Single-blind, Randomised, Placebo Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK1034702 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of GSK1034702 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 110623
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cognitive Disorders
Keywords: schizophrenia; M1 receptor agonist; safety; pharmacokinetics; GSK1034702
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia | interventions — GSK 1034702

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Other): Subjects will be receive GSK1034702 0.5 milligram (mg) following the dose escalation plan
  Interventions: Drug: GSK1034702; Drug: Placebo
- Cohort 2 (Other): Subjects will be receive GSK1034702 5 mg following the dose escalation plan
  Interventions: Drug: GSK1034702; Drug: Placebo

INTERVENTIONS:
Drug: GSK1034702 — Oral or liquid
Drug: Placebo — To match GSK1034702

SUMMARY:
This is a First Time in Human Study to assess the safety, tolerability and pharmacokinetics of single doses of GSK1034702 in healthy subjects. It will be a single-blind, randomized, placebo-controlled, single oral dose, dose-rising, cross-over study in healthy male and female (of non-child bearing potential) subjects. Subjects will be randomized into cohorts of 10 subjects and cohorts will be recruited until the pre-defined safety or PK stopping limits are reached. Each subject will receive placebo and up to 4 doses of GSK1034702 in a randomized sequence on 5 separate study occasions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including own and familial medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 55 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential
* Body weight > 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Capable of reading, comprehending and writing English at a sufficient level to complete study-related materials.
* Demonstrates no evidence of mental impairment.
* No co-morbid Psychiatric Disorders as defined using the Mini International Neuropsychiatric Interview

Exclusion Criteria:

* A positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B , Hepatitis C or HIV.
* History of regular alcohol consumption.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements .
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females, females planning pregnancy or lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects with a current or a history of psychiatric illness.
* Subjects with any history of suicidal attempts or behavior.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice (and pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices) from 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05-02 (Actual); Primary Completion 2008-12-15 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
•Safety and tolerability determined by adverse events; ECG; Holter; blood pressure, heart rate, respiration rate; clinical laboratory evaluations, pupil size & temperature.•Blood concentrations of GSK1034702. | 20 weeks

SECONDARY OUTCOMES:
Assessment of the Bond-Lader Visual Analogue Scale. | 20 weeks
Assessment of exploratory PD markers: neuroendocrine markers, e.g. growth hormone. | 20 weeks
Relationship between GSK1034702 plasma concentrations and safety/tolerability or exploratory PD endpoints with selected pharmacodynamic and safety parameters. | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 110623 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/110623?search=study&search_terms=110623#rs